CLINICAL TRIAL: NCT00610727
Title: Tolerability, Safety and Pharmacokinetics of a Single Dose of Staccato™ Prochlorperazine for Inhalation in Normal, Healthy Volunteers
Brief Title: Staccato Prochlorperazine Single Dose PK Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-004-001
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Migraine
Keywords: Migraine, Prochlorperazine aerosol
MeSH Terms: conditions — Migraine Disorders | interventions — Prochlorperazine

STUDY DESIGN:
Intervention Model Description: Stage 1: open-label, single-dose stage with 3 treatment periods divided into 2 phases Stage 2: double-blind, placebo-controlled, dose-escalation treatment period
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Stage 2 was a double-blind, placebo-controlled, 4 step dose-escalation trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Inhaled prochlorperazine 0.625 mg vs IV (Experimental): Prochlorperazine 0.5 mg IV over 5 sec crossover Inhaled prochlorperazine 0.625 mg
  Interventions: Drug: Prochlorperazine 0.5 mg IV over 5 sec; Drug: Inhaled prochlorperazine 0.625 mg; Drug: Prochlorperazine 10 mg IV over 5 sec
- Inhaled prochlorperazine 1.25 mg (Experimental): Inhaled Staccato prochlorperazine 1.25 mg
  Interventions: Drug: Inhaled prochlorperazine 1.25 mg
- Inhaled prochlorperazine 2.5 mg (Experimental): Inhaled Staccato prochlorperazine 2.5 mg
  Interventions: Drug: Inhaled prochlorperazine 2.5 mg
- Inhaled prochlorperazine 5 mg (Experimental): Inhaled Staccato prochlorperazine 5 mg
  Interventions: Drug: Inhaled prochlorperazine 5 mg
- Inhaled prochlorperazine 10 mg (Experimental): Inhaled Staccato prochlorperazine 10 mg
  Interventions: Drug: Inhaled prochlorperazine 10 mg
- inhaled Placebo (Placebo Comparator): inhaled Staccato Placebo (0 mg)
  Interventions: Drug: Inhaled placebo

INTERVENTIONS:
Drug: Prochlorperazine 0.5 mg IV over 5 sec — IV Prochlorperazine for bioavailability
  Other Names: PCZ
  Arms: Inhaled prochlorperazine 0.625 mg vs IV
Drug: Inhaled prochlorperazine 0.625 mg — Inhaled Staccato Prochlorperazine 0.625 mg
  Other Names: PCZ
  Arms: Inhaled prochlorperazine 0.625 mg vs IV
Drug: Inhaled prochlorperazine 1.25 mg — Inhaled Staccato Prochlorperazine 1.25 mg
  Other Names: PCZ
  Arms: Inhaled prochlorperazine 1.25 mg
Drug: Inhaled prochlorperazine 2.5 mg — Inhaled Staccato Prochlorperazine 2.5 mg
  Other Names: PCZ
  Arms: Inhaled prochlorperazine 2.5 mg
Drug: Inhaled prochlorperazine 5 mg — InhaledStaccato Prochlorperazine 5 mg
  Other Names: PCZ
  Arms: Inhaled prochlorperazine 5 mg
Drug: Inhaled prochlorperazine 10 mg — InhaledStaccato Prochlorperazine 10 mg
  Other Names: PCZ
  Arms: Inhaled prochlorperazine 10 mg
Drug: Inhaled placebo — Inhaled Staccato Placebo (0 mg)
  Other Names: ADASUVE placebo
  Arms: inhaled Placebo
Drug: Prochlorperazine 10 mg IV over 5 sec — Prochlorperazine 10 mg IV over 5 sec for patient qualification
  Other Names: PCZ
  Arms: Inhaled prochlorperazine 0.625 mg vs IV

SUMMARY:
The objective of this study was to evaluate the tolerability, safety, and pharmacokinetics of inhaled prochlorperazine

DETAILED DESCRIPTION:
The objective of this study was to evaluate the tolerability, safety, and pharmacokinetics of a single, inhaled dose of prochlorperazine (PCZ), administered as 1 or 2 puffs in healthy young volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be male or female subjects between the ages 18 to 45 years, inclusive in good general health as determined by medical history, physical examination, 12-lead ECG, spirometry, blood chemistry profile, hematology, urinalysis and in the opinion of the Principal Investigator.

Exclusion Criteria:

* Subjects with a known history of allergy or intolerance to phenothiazines or related drugs or who have any disease, by history, physical examination, or laboratory abnormalities that in the investigator's opinion, would present undue risk to the subject, or may confound the interpretation of study results.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2004-08; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Spyker, MD, Study Director — Alexza Pharmaceuticals, Inc.
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

REFERENCES:
- [Background] Avram MJ, Spyker DA, Henthorn TK, Cassella JV. The pharmacokinetics and bioavailability of prochlorperazine delivered as a thermally generated aerosol in a single breath to volunteers. Clin Pharmacol Ther. 2009 Jan;85(1):71-7. doi: 10.1038/clpt.2008.184. Epub 2008 Oct 1. PMID 18830225

RESULTS

PARTICIPANT FLOW:
Groups:
- Qualification & Crossover Arm, Inhaled Prochlorperazine vs IV: Prochlorperazine 10 mg IV over 2 min qualification
  Prochlorperazine 0.5 mg IV over 5 sec crossover Inhaled prochlorperazine 0.625 mg
  ALL SUBJECTS RECEIVED ALL TREATMENT
Period: Overall Study
Arm/Group | Qualification & Crossover Arm, Inhaled Prochlorperazine vs IV | Inhaled Prochlorperazine 1.25 mg | Inhaled Prochlorperazine 2.5 mg | Inhaled Prochlorperazine 5 mg | Inhaled Prochlorperazine 10 mg | Inhaled Placebo
Started | 14 | 8 | 8 | 8 | 8 | 8
Completed | 14 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Qualification & Crossover, Inhaled Prochlorperazine vs IV: Prochlorperazine 10 mg IV over 2 min qualification
  Prochlorperazine 0.5 mg IV over 5 sec crossover Inhaled prochlorperazine 0.625 mg
  ALL SUBJECTS RECEIVED ALL 3 TREATMENTS
- Total: Total of all reporting groups
Arm/Group | Qualification & Crossover, Inhaled Prochlorperazine vs IV | Inhaled Prochlorperazine 1.25 mg | Inhaled Prochlorperazine 2.5 mg | Inhaled Prochlorperazine 5 mg | Inhaled Prochlorperazine 10 mg | Inhaled Placebo | Total
Number analyzed (Participants) | 14 | 8 | 8 | 8 | 8 | 8 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 8 | 8 | 8 | 8 | 8 | 54
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (7.86) | 25.1 (3.44) | 25 (4.57) | 26.4 (8.94) | 28.8 (10.2) | 23.5 (7.03) | 25.8 (7.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 4 | 4 | 4 | 4 | 26
  Male | 8 | 4 | 4 | 4 | 4 | 4 | 28
Region of Enrollment [Number; unit: participants]
  United States | 14 | 8 | 8 | 8 | 8 | 8 | 54

OUTCOME MEASURES:

1. Primary Outcome: Time to Peak (Tmax)
Description: Time from dose to peak prochlorperazine concentration
Time Frame: 24 hours
Population: Pharmacokinetic Population
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- 0.5 mg 5 Sec IV: 0.5 mg 5 sec IV prochlorperazine
- 0.625 mg Inhaled Prochlorperazine: 0.625 mg Inhaled prochlorperazine drug
- 1.25 mg Inhaled: 1.25 mg Inhaled Prochlorperazine
- 2.5 mg Inhaled: 2.5 mg Inhaled Prochlorperazine
- 5 mg Inhaled: 5 mg Inhaled Prochlorperazine
- 10 mg Inhaled: 10 mg Inhaled Prochlorperazine
Arm/Group | 0.5 mg 5 Sec IV | 0.625 mg Inhaled Prochlorperazine | 1.25 mg Inhaled | 2.5 mg Inhaled | 5 mg Inhaled | 10 mg Inhaled
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 8 | 8
hours | 0.042 [0.025 to 0.067] | 0.033 [0.025 to 0.042] | 0.025 [0.013 to 0.082] | 0.033 [0.017 to 0.033] | 0.040 [0.017 to 0.115] | 0.033 [0.013 to 0.108]

2. Secondary Outcome: Absolute Bioavailability of Inhaled Prochlorperazine
Description: Absolute bioavailability of inhaled prochlorperazine via AUC infinity
Time Frame: 24 hours
Population: Bioavailability crossover subjects, n=8
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Fraction absorbed
Groups:
- Bioavailability Crossover Arm: 0.625 mg prochlorperazine crossover 0.5 mg via 5-second IV prochlorperazine
Arm/Group | Bioavailability Crossover Arm
Number analyzed (Participants) | 8
Fraction absorbed | 0.98 [0.73 to 1.34]

3. Secondary Outcome: Dose Proportionality of Inhaled Prochlorperazine by Power Analysis
Description: Dose proportionality by power analysis examines the linear regression of the log-AUC versus log-Dose on a by-patient basis across all doses administered. The slope and 90% confidence interval (CI) provide a clear, quantitative (best practices) assessment of the relationship of drug delivered to dose administered. The units on such analyses are generally those of slope (rise over run), with 1.000 being "perfect". Although any positive slope might be considered clinically useful, a 90% CI within the criteria of 0.800-1.250 may be considered a delivery system which is "as good as it gets".
Time Frame: 24 hours
Population: Pharmacokinetic Population, n=40
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Slope of Power Regression
Groups:
- All Subjects Receiving Inhaled Prochloperazine: 0.625 mg, 8 subjects 1.25 mg, 8 subjects 2.5 mg, 8 subjects 5 mg, 8 subjects 10 mg, 8 subjects
Arm/Group | All Subjects Receiving Inhaled Prochloperazine
Number analyzed (Participants) | 40
Slope of Power Regression | 1.089 [.99 to 1.2]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were considered treatment related from the first exposure to study treatment until 30 days after the last treatment
Description: Adverse events (AEs) were assessed predose and Performed throughout the 24-hour period after dosing .
Groups:
- IV Prochlorperazine 10 mg: Intravenous prochlorperazine 10 mg
- IV Prochlorperazine 0.5 mg: Intravenous prochlorperazine 0.5 mg
- Inhaled Prochlorperazine 0.625: Inhaled prochlorperazine 0.625 mg
Arm/Group | IV Prochlorperazine 10 mg | IV Prochlorperazine 0.5 mg | Inhaled Prochlorperazine 0.625 | Inhaled Prochlorperazine 1.25 mg | Inhaled Prochlorperazine 2.5 mg | Inhaled Prochlorperazine 5 mg | Inhaled Prochlorperazine 10 mg | Inhaled Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 6/14 | 0/8 | 0/8 | 5/8 | 3/8 | 0/8 | 4/8 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Prochlorperazine 10 mg (N=14) | IV Prochlorperazine 0.5 mg (N=8) | Inhaled Prochlorperazine 0.625 (N=8) | Inhaled Prochlorperazine 1.25 mg (N=8) | Inhaled Prochlorperazine 2.5 mg (N=8) | Inhaled Prochlorperazine 5 mg (N=8) | Inhaled Prochlorperazine 10 mg (N=8) | Inhaled Placebo (N=8)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sensation of pressure in face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less